CLINICAL TRIAL: NCT01260129
Title: Safety and Efficacy of 8mg Once-daily Versus 4mg Twice-daily Silodosin With Lower Urinary Tract Symptoms Suggestive of BPH ; 12-week, Double-blind, Randomized, Comparison, Multi-center Study
Brief Title: Safety and Efficacy of QD Versus BID Silodosin With Lower Urinary Tract Symptoms Suggestive of BPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CWP-SDS-401
Record Dates: First submitted 2010-10-28; First posted 2010-12-15 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Benign Prostatic Hypertrophy
Keywords: BPH; silodosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — silodosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Silodosin 8 mg (Experimental)
  Interventions: Drug: Silodosin
- Silodosin 4 mg (Experimental)
  Interventions: Drug: Silodosin

INTERVENTIONS:
Drug: Silodosin — Silodosin 8 mg orally, once daily after morning meal
  Arms: Silodosin 8 mg
Drug: Silodosin — Silodosin 4 mg orally, twice daily after morning and evening meal
  Arms: Silodosin 4 mg

SUMMARY:
Korea has newly adopted 8mg Silodosin once daily. Against these backdrops, this clinical study is designed to demonstrate that the newly adopted dose is not inferior to the existing dose in its efficacy and safety.

DETAILED DESCRIPTION:
Silodosin is a highly selective α1A-adrenoceptor antagonist for the treatment of the signs and symptoms of BPH. 4mg Silodosin twice daily has been approved in Asia including Japan and Korea. In US, 8mg Silodosin once daily with the FDA approval is already available. Korea has newly adopted 8mg Silodosin once daily. Against these backdrops, this clinical study is designed to demonstrate that the newly adopted dose is not inferior to the existing dose in its efficacy and safety. The study used double-blind, random assignment in Korean men with signs and symptoms of BPH for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

Patients who have been diagnosed with BPH through digital rectal exam or ultrasonographic findings and meet the following criteria.

* Outpatients aged 50 or over
* Patients with a total I-PSS score of 8 or higher and a QoL score of 3 or higher
* Patients with a prostate volume measured by transabdominal ultrasonography, or TRUS of 20 ml or greater
* Patients with a maximum urinary flow rate (Qmax_) of 15ml/sec or below (whose a void urinary volume of 120ml or greater)

Exclusion Criteria:

* Patients with a residual urinary volume of 200ml or greater
* Patients with a history of prostatectomy
* Patients with a history of intrapelvic radiation therapy
* Patients with a history of prostatic hyperthermia
* Patients with prostate cancer or suspected prostate cancer
* Patients with complications considered likely to affect urinary passing such as neurogenic bladder, bladder calculus and active urinary tract infection. UTI
* Patients conducting self-catheterization
* Patients with renal impairment (serum creatinine of 3.0 mg/dl or greater)
* Patients with severe heptic disorders (hepatic insufficiency, cirrhosis, jaundice, hepatoma) or with a total bilirubin of 3.0mg/dL or greater or AST/ALT 2.5 times higher than normal level
* Patients with history of severe arrhythmia, cardiac failure, cardiac infarction, unstable angina, cerebral infarction within 6 months
* Patients with a history of an allergy to α-blockers
* Patients with orthostatic hypotension at around screening visit
* Patients with an experience of other investigational product treatments within 4 weeks form screening visit.
* Patients with a PSA of 10 or over, Patients with tumor identified by a prostate biopsy with a PSA of 4 or over (For patients taking 5α-reductase inhibitors for more than 3 months are presumed to have double than their actual PSA levels.)
* Patients who have taken unstable doses of antidepressants within the 3 months or who are expected to take unstable doses during the study
* Patients who have taken alpha blockers within the 2 weeks from the start of the therapy
* Patients who have taken unstable doses of 5α-reductase inhibitors within the 3 months from the start of the therapy or who are expected to take unstable doses during the study.
* Patients disqualified by the investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
I-PSS | 12 weeks
  Change in I-PSS total score from baseline

SECONDARY OUTCOMES:
I-PSS, Qmax, QoL, ICS Male Questionnaire, goal achievement, Treatment satisfaction question | 12 weeks
  * The rate of patients who experience a decrease in I-PSS total score of 25% or higher
  * The rate of patients who experience an improvement of at least 4 in I-PSS total score I-PSS
  * Change in Qmax from baseline
  * The rate of patients who experience an improvement of 30% or over in Qmax
  * Change in the I-PSS voiding and storage scores from baseline
  * Change in QoL score from baseline
  * Change in ICS Male Questionnaire from baseline
  * Patient's goal achievement score
  * Treatment Satisfaction Question

CONTACTS AND LOCATIONS:
Overall Officials: Jae Seung Paick, ph.D, Principal Investigator — Department of Urology, Seoul National University Hospital
Locations (14):
- South Korea (14):
  - The Catholic Univ., Bucheon ST.Mary's Hospital, Bucheon-si
  - Busan National Univ. Hospital, Busan
  - Konkuk Univ, Chungju Hospital, Chungju
  - Choongnam National Univ. Hospital, Daejeon
  - Eulji Univ. Hospital, Daejeon
  - Chonnam Univ. Hospital, Hwasun
  - Inha Univ. Hosipital, Incheon
  - Asan Medical Center, Seoul
  - Chungang Univ. Hospital, Seoul
  - Korea Univ. Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic Univ., Seoul ST.Mary's Hospital, Seoul